CLINICAL TRIAL: NCT05884346
Title: Association Between Coronary and Peripheral Vascular Injury in Heart Failure Patients With Preserved Ejection Fraction.
Acronym: COROVASC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP230214; 2022-A02455-38 (Other: Agence Nationale de Sécurité du Médicament et des produits de santé); 23.00664.000175 (Other: Commission Nationale des Recherche Impliquant la Personne Humaine)
Record Dates: First submitted 2023-05-10; First posted 2023-06-01 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Ultrahigh-frequency ultrasound; Heart Failure with Preserved Ejection Fraction; Microcirculation; Arterial remodeling; Small arteries; Ischemia
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heart Failure Preserved Ejection Fraction with coronary disease (Other)
  Interventions: Other: Ultrahigh-frequency ultrasound
- Heart Failure Preserved Ejection Fraction without coronary disease (Other)
  Interventions: Other: Ultrahigh-frequency ultrasound

INTERVENTIONS:
Other: Ultrahigh-frequency ultrasound — Arterial remodeling of the digital arteries will be measured by ultrahigh-frequency ultrasound and will be compared in heart failure patients with preserved ejection fraction with and without identified macroscopic coronary disease

SUMMARY:
Heart failure with preserved ejection fraction (HPEF, defined as LVEF ≥50%) represents 50% of hospital admissions for heart failure. Although its morbi-mortality is similar to that of heart failure with reduced ejection fraction (HFPEF), it remains an unknown disease with limited data especially from an etiological point of view. The underlying causes are imperfectly understood, and more than half of the patients have HPEF labeled "idiopathic."

A non-hierarchical clustering study of HPEF patients led to the identification of a subgroup of patients (25%) with a predominant coronary vascular phenotype (i.e., a history of coronary stenosis with or without the need for revascularization). In these patients, vascular endothelial dysfunction would play a central role in the development and progression of heart failure.One of the mechanisms leading to HPEF could be a decrease in the bioavailability of nitric oxide (NO) involved in the relaxation of the cardiac muscle. As the mechanism of action of NO is pleiotropic, a decrease in NO bioavailability could also be observed at the peripheral level, favoring in the long term the development of unfavorable vascular remodeling, for example in the small digital or retinal arteries.Some HPEF patients could thus be distinguished from others by their predominant "vascular" profile. The link between HPEF and endothelial dysfunction has been suspected but never clearly demonstrated.

Ultra-high frequency ultrasound is an innovative technology to estimate the remodeling of small distal arteries in a non-invasive way. The investigators propose to use this imaging on digital arteries in HPEF patients and to study the association with known coronary macrovascular damage.The remodeling parameters will be measured and compared in patients with HPEF with or without identified macrovascular coronary disease.This characterization of arterial remodeling on the digital arteries could be a powerful tool for non-invasive screening in the identification of a subgroup of HPEF that is still considered idiopathic.

ELIGIBILITY:
Inclusion Criteria :

Group 1 :

* Patients who are ≥ 18 years old
* Heart failure with preserved ejection fraction (LVEF ≥ 50%)
* B-type natriuretic peptide (BNP) > 35 pg/mL at inclusion
* Coronary macrovascular disease (significant coronary stenosis, which may have required revascularization by stenting or coronary bypass surgery).

Group 2 :

* Patients who are ≥ 18 years old
* Heart failure with preserved ejection fraction (LVEF ≥ 50%)
* B-type natriuretic peptide (BNP) > 35 pg/mL at screening
* Absence of coronary macrovascular disease (no significant coronary atheroma (< 30%) or history of stenting or coronary bypass surgery).

Non-inclusion Criteria :

Group 1 and group 2 :

* Patients under legal protection
* Patients not affiliated to a Social Security system
* Patient under State Medical Help (France - AME)
* Pregnancy or breastfeeding
* Refusal or inability to sign consent
* Known and treated retinal vasculopathy
* Severe or non-stabilized hypertension (BP > 180/100 mmHg at screening)
* History of LVEF < 40%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Digital vascular remodeling by ultrahigh-frequency ultrasound | Day 1
  The wall-to-lumen ratio of digital arteries recorded with ultrahigh-frequency ultrasound.

SECONDARY OUTCOMES:
Radial vascular remodeling by echo-tracking | Day 1
  Measurement of peripheral vascular remodeling on radial arteries by arterial distension parameters.
Carotid vascular remodeling by echo-tracking | Day 1
  Measurement of peripheral vascular remodeling on carotid arteries by arterial distension parameters.
Endothelial dysfunction | Day 1
  Level of endothelial function measured by arterial flow-mediated vasodilation (FMD, expressed in %).
Pulse wave velocity | Day 1
  Pulse wave velocity (PWV, velocity expressed in m/s) carotid-femoral (aortic elasticity).
Retinal microvascularization | Day 1
  To study the retinal microvascularization by Optical Coherence Tomography Angiography (OCT-A) : density measurement per sector (% per studied area).
Calcium score | Day 1
  Compare the calcium score (expressed by the Agatston score) in patients with heart failure with preserved ejection fraction with or without a priori coronary artery disease.

CONTACTS AND LOCATIONS:
Overall Officials: Roxane GAÏSSET, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital européen Georges Pompidou - AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: No